CLINICAL TRIAL: NCT02668276
Title: The Impact of a Gene Expression Profile on Treatment Choice and Outcome Among Minority Men Newly Diagnosed With Prostate Cancer: A Randomized Trial
Brief Title: Engaging Newly Diagnosed Men About Cancer Treatment Options
Acronym: ENACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Cook County Hospital (Other); Genomic Health®, Inc. (Industry)
Responsible Party: Principal Investigator, Peter Gann, Professor of Pathology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-1294; W81XWH-14-PCRP-BDA (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; Oncotype DX; Treatment Decisions
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard NCCN counseling (Placebo Comparator): National Comprehensive Cancer Network (NCCN) counseling uses recommendations based on currently-accepted approaches to cancer treatment.
  Interventions: Other: Standard NCCN counseling
- Standard NCCN counseling and Oncotype DX results (Experimental): National Comprehensive Cancer Network (NCCN) counseling uses recommendations based on currently-accepted approaches to cancer treatment. The result provided by the Oncotype DX prostate test is called a Genomic Prostate Score (GPS). The GPS provides important information about how aggressive a man's cancer is based on the biology of the man's individual tumor.
  Interventions: Other: Standard NCCN counseling and Oncotype DX results

INTERVENTIONS:
Other: Standard NCCN counseling
  Arms: Standard NCCN counseling
Other: Standard NCCN counseling and Oncotype DX results
  Arms: Standard NCCN counseling and Oncotype DX results

SUMMARY:
This research is being done to better understand how a new lab test called the Oncotype DX Prostate Cancer Assay may impact what treatment men decide to get and how they feel and think about their choice of treatment. The study will compare men who receive this new lab test with men who receive the usual counseling given to men after they get a new diagnosis of prostate cancer. Prostate cancer is sometimes slow-growing and sometimes fast-growing. Healthcare providers are searching for better ways to predict how each tumor will behave so that each man can make a better decision about when to receive treatment. The Oncotype DX lab test uses leftover prostate biopsy tissue to generate a Genomic Prostate Score (GPS). The GPS is related to the risk of a fast-growing cancer being discovered if surgery is performed to remove a man's prostate. The goal of this study is to find out if this test helps men when they are deciding how their prostate cancer will be treated. Treatment options include surgery to remove the prostate, radiation therapy, or an approach called "active surveillance" in which there is no immediate therapy and the tumor is watched using prostate specific antigen (PSA) tests and repeat biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Men with newly diagnosed prostate cancer who are categorized as Very Low, Low, or Intermediate risk by NCCN criteria;
* Are age 76 or younger

Exclusion Criteria:

* Men who are categorized as High or Very High risk by NCCN criteria;
* Men who have already received counseling from their urologist about their treatment options and have decided to undergo treatment, active surveillance, or watchful waiting;
* Men age 77 or older

Max Age: 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Effect of adding Oncotype DX prostate cancer assay to usual counseling on the proportion of men adopting Active Surveillance (AS). | 3-6 months after treatment decision

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Gann, MD, ScD, Principal Investigator — University of Illinois at Chicago; Adam B Murphy, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Jesse Brown V. A. Medical Center, Chicago, Illinois
  - John H. Stroger Hospital of Cook County, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Murphy AB, Abern MR, Liu L, Wang H, Hollowell CMP, Sharifi R, Vidal P, Kajdacsy-Balla A, Sekosan M, Ferrer K, Wu S, Gallegos M, King-Lee P, Sharp LK, Ferrans CE, Gann PH. Impact of a Genomic Test on Treatment Decision in a Predominantly African American Population With Favorable-Risk Prostate Cancer: A Randomized Trial. J Clin Oncol. 2021 May 20;39(15):1660-1670. doi: 10.1200/JCO.20.02997. Epub 2021 Apr 9. PMID 33835822